CLINICAL TRIAL: NCT00327106
Title: Efficacy of Tranexamic Acid on Perioperative Blood Loss During Hip Fracture Surgery.
Brief Title: Tranexamic Acid in HIp Fracture Surgery (THIF Study)
Acronym: THIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, Centre Hospitalier Universitaire de Saint-Etienne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0401129; DGS 2005-01094
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Hip Fracture
Keywords: hip fracture; transfusion; tranexamic acid; fondaparinux
MeSH Terms: conditions — Hip Fractures | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Exacyl
  Interventions: Drug: Tranexamic acid (Exacyl)
- 2 (Placebo Comparator): Physiologic serum
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid (Exacyl) — 15 mg/kg IV (in the vein), just before surgery and 3 hours after surgery
  Other Names: Exacyl
  Arms: 1
Drug: Placebo — NaCl 9‰, 0,15 ml/kg IV (in the vein), just before surgery and 3 hours after surgery.
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy of tranexamic acid in hip fracture surgery on the reduction of allogeneic red blood cell transfusion.

DETAILED DESCRIPTION:
Studies in hip and knee arthroplasty (scheduled surgery) have shown that tranexamic acid decreases allogeneic red blood cell transfusion. In hip fracture surgery, an emergent procedure, transfusion is frequent. Transfusion increases adverse events such as postoperative bacterial infection and venous thrombosis. The purpose of this study is to assess the efficacy of tranexamic acid, an anti-fibrinolytic agent, in hip fracture surgery on the reduction of allogeneic red blood cell transfusion. The trial will also evaluate if the reduction in transfusion will be associated with less postoperative infection and without an increase in the thrombotic risk.

Patients with an isolated hip fracture of less than 48 hours will be randomized to either tranexamic acid 15mg/kg IV at skin incision and three hours later or saline.Patients will receive fondaparinux for prophylaxis of venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring surgery for an isolated hip fracture of less than 48 hours

Exclusion Criteria:

* Contraindication to tranexamic acid
* Contraindication to fondaparinux
* Contraindication to general anesthesia associated with a femoral nerve block
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
number of patients receiving the transfusion of at least one unit of allogeneic red blood cell | between the begining of surgery (day 1) and the eighth post-operative day (day 8)

SECONDARY OUTCOMES:
number of patients receiving the transfusion of at least one unit of allogeneic red blood cell | between the administration of fondaparinux for venous thrombosis prophylaxis(8 hours after end of surgery on day 1) and the eighth post-operative day (day 8)
post-operative major hemorrhage | day 8
post-operative blood loss | untill day 8
post-operative bacterial infection (combined criteria of wound infection, bronchopulmonary infection and urinary tract infection) | untill six weeks
thromboembolic events (combined criteria of venous thrombo-embolism, stroke, acute coronary syndrome and peripheral arterial thrombosis) | untill six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Zufferey, Doctor, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Étienne-de-Montluc, Pays de la Loire Region, France

REFERENCES:
- [Derived] Zufferey PJ, Miquet M, Quenet S, Martin P, Adam P, Albaladejo P, Mismetti P, Molliex S; tranexamic acid in hip-fracture surgery (THIF) study. Tranexamic acid in hip fracture surgery: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):23-30. doi: 10.1093/bja/aep314. PMID 19926634